CLINICAL TRIAL: NCT01257659
Title: STARR Type Trans-anal Resection Versus Vaginal Rectocele Repair Using a Posterier Elevate Prothesis: a Randomized, Multicentric, Prospective Study on Defecatory Function
Brief Title: STARR Trans-anal Resection Versus Vaginal Rectocele Repair Using Elevate: Effects on Defecatory Function
Acronym: RectoVerso
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find enough patients who accept randomization of surgical procedures.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC-I/2010/RdeT-01; 2010-A00665-34 (Other: Agence Française de Sécurité Sanitaire des Produits de Santé (Afssaps))
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Rectocele
Keywords: Rectocele; Trans anal STARR resection; Transvaginal repair
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STARR arm (Experimental): In this group of patients, the STARR transanal stapling system is used to treat the rectocele.
  Interventions: Procedure: STARR rectocele repair
- Elevate arm (Active Comparator): In this group of patients, a posterior Elevate mesh is placed transvaginally to treat the rectocele.
  Interventions: Procedure: Elevate mesh rectocele repair

INTERVENTIONS:
Procedure: STARR rectocele repair — The STARR transanal stapling system is used to repair a rectocele.
  Arms: STARR arm
Procedure: Elevate mesh rectocele repair — A posterior Elevate mesh is placed transvaginally to repair a rectocele.
  Arms: Elevate arm

SUMMARY:
The primary objective of this study is to compare the function results between two methods for surgically repairing rectoceles: vaginal versus endo-anal surgery. Our working hypothesis is that the relatively new type of endo-anal surgery will result in better voiding function compared to the traditional vaginal surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient is not under any type of guardianship
* patient has a rectocele > 3 cm during defecography
* patient has persistent defecatory troubles depite medical treatment (laxatives for at least 1 month) and an ODS score > 10
* patient recieved information and signed the consent form

Exclusion Criteria:

* patient cannot read French
* patient has an asymptomatic rectocele
* patient with an enterocele at rest upon defecography, with opacification of the small bowel
* patient with non-rehabilitated anorectal asynchrony (anism)
* patient with anal incontinence, Wexner score > 7
* patient has a rectal lesion
* patient has previously had rectal surgery including a colorectal anastomosis
* patient has previously had a surgery involving disection of the rectovaginal wall, except for myorraphy of relever muscles
* patient has previously had pelvic radiotherapy
* anal sphincter insufficiency detected by rectomanometry
* megarectum detected by rectomanometry and defecography
* granule transit anomaly: > 70h
* exteriorized rectal prolapse
* rectovaginal fistule
* intestinal inflammatory disease
* anal stenosis
* anal or rectal tumor
* patient refuses to participate or refuses to sign consent
* patient is enrolled in another study
* contra indication for general or localized anesthesia
* patient does not have social security coverage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
presence/absence of a 50% drop in the ODS score | 12 months
  presence/absence of a 50% drop in the ODS score: constipation score defined by Altomare et al, 2008.

SECONDARY OUTCOMES:
presence/absence of prolapse recurrence | 6 weeks
  presence/absence of prolapse recurrence: determined by prolapse staging
Frequency of laxative use | 6 weeks
Intervention time (min) | 1 day
Questionnaire PFDI 20 | 6 weeks
Questionnaire PFIQ 7 | 6 weeks
Questionnaire SF 36 | 6 weeks
Questionnaire PISQ-12 | 6 weeks
presence/absence of prolapse recurrence | 6 months
  presence/absence of prolapse recurrence: determined by prolapse staging
presence/absence of prolapse recurrence | 12 months
  presence/absence of prolapse recurrence: determined by prolapse staging
presence/absence of prolapse recurrence | 36 months
  presence/absence of prolapse recurrence: determined by prolapse staging
Frequency of laxative use | 6 months
Frequency of laxative use | 12 months
Frequency of laxative use | 36 months
Questionnaire PFDI 20 | 6 months
Questionnaire PFDI 20 | 12 months
Questionnaire PFDI 20 | 36 months
Questionnaire PFIQ 7 | 6 months
Questionnaire PFIQ 7 | 12 months
Questionnaire PFIQ 7 | 36 months
Questionnaire SF 36 | 6 months
Questionnaire SF 36 | 12 months
Questionnaire SF 36 | 36 months
Questionnaire PISQ-12 | 6 months
Questionnaire PISQ-12 | 12 months
Questionnaire PISQ-12 | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Renaud de Tayrac, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - Hôpital de la Conception, Marseille
  - Clinique Beau Soleil, Montpellier
  - Clinique Adassa, Strasbourg
  - Hôpital Paule de Viguier, CHU de Toulouse, Toulouse
  - Hôpital Purpan, CHU de Toulouse, Toulouse